CLINICAL TRIAL: NCT04073901
Title: Clinical Evaluation of Endocrowns Versus Prefabricated Zirconia Crowns in Pulpotomized Primary Molars : A Pilot Prospective Clinical Study
Brief Title: Comparative Study Between Zirconia Crowns and Endocrowns in Pulpotomized Primary Molars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nahda University (Other)
Responsible Party: Principal Investigator, Yassmine mohamed farouk el makawi, Assistant lecturer, Minia University
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 186
Record Dates: First submitted 2019-08-22; First posted 2019-08-29 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Paediatric; Dentistry
Keywords: Aesthetic; Endo-crowns; primary; molars; pulpotomy; zirconium; crowns

STUDY DESIGN:
Masking Description: only satiation was blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endocrown (Experimental): Adhesive monoblock restoration for pulpotomized primary molars
  Interventions: Other: Endocrowns
- Zirconia crowns (Active Comparator): Prefabricated primary full coverage crown
  Interventions: Other: Endocrowns

INTERVENTIONS:
Other: Endocrowns — Adhesive monoblock restoration for pulpotomized primary molars

SUMMARY:
Objectives: The new approach of pediatric esthetic dentistry intended to achieve a healthy beautiful smile rather than achieving only a beautiful smile. The objective of this study was to assess the clinical performance of ceramic Endocrowns and Zirconia crowns for the restoration of pulpotomized primary molars and parental satisfaction toward these crowns. Study design: Randomized clinical trial/split mouth design compared the clinical outcomes of two coronal restorations, on patients with bilateral carious second primary molars restoring one side with Endocrown (IPS e.max Press) and the other side with zirconia crown. Children attended Nahda University; Faculty of Dentistry clinics who need restorations screened for inclusion criteria till 20 patients are recruited (20 teeth for zirconia crown restorations and 20 for Endocrowns restorations). All children fulfilled the inclusion criteria were evaluated for factors including restoration integrity, marginal adaptation, marginal discoloration, oral health and overall clinical success at 3,6,12 months while parental satisfaction at 12 months follow up..

ELIGIBILITY:
Inclusion Criteria:

1. . Free of systemic diseases.
2. Age between 4 and 7 years.
3. Takes no medication on regular basis.
4. Has bilateral lower second primary molar with deep carious lesion, indicated for pulp therapy and crown restoration. (split mouth)
5. Patient and parent compliance.

Exclusion Criteria:

* 1. Non-restorable tooth. 2. Tooth near its exfoliation. 3. Tooth with extensive root resorption or periapical pathosis.

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Enrollment: 20 (Actual)
Dates: Start 2018-02-02 (Actual); Primary Completion 2018-06-03 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Restoration integrity | one year
  Modified USPHS(United States Public Health Service (USPHS), alpha criteria rating system)
marginal adaptation | one year
  Modified USPHS(United States Public Health Service (USPHS), alpha criteria rating system)
marginal discoloration | one year
  Modified USPHS(United States Public Health Service (USPHS), alpha criteria rating system)

SECONDARY OUTCOMES:
parent satisfaction | immediate after intervention
  5-point Likert scale Likert scale(0-4)

CONTACTS AND LOCATIONS:
Locations (1):
- Yassmine Mohamed Farouk El Makawi, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No